CLINICAL TRIAL: NCT07307378
Title: Evaluation of Lower Limb Biomechanical Analysis of Roundhouse Kick in Elite and Youth Taekwondo Athletes Through Functional Principal Component Analysis.
Brief Title: Lower Limb Biomechanics of the Roundhouse Kick in Elite and Youth Taekwondo Athletes Using FPCA
Status: Active, not recruiting | Type: Observational
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Shazlin Shaharudin, Associate Professor, School of Health Sciences, Universiti Sains Malaysia, Universiti Sains Malaysia
Other Study IDs: USM/JEPeM/KK/25030312
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Taekwondo Roundhouse Kick Biomechanics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Youth Taekwondo Athletes: Youth taekwondo athletes who will complete one laboratory testing session (roundhouse kick trials) for motion analysis and surface EMG. No intervention.
- Elite Taekwondo Athletes: Elite taekwondo athletes who will complete one laboratory testing session (roundhouse kick trials) for motion analysis and surface EMG. No intervention.

SUMMARY:
This study aims to understand how the lower limbs (hip, knee, and ankle) function during a taekwondo roundhouse kick. Elite and youth taekwondo athletes will be compared to identify movement and muscle-activation patterns related to kicking performance. Participants will attend one testing session at Ludong University, China. During the session, participants will complete a standardized warm-up and then perform a series of roundhouse kicks. Body movement will be recorded using motion-analysis equipment, and muscle activity will be recorded using surface electromyography (EMG) sensors placed on the skin. These recordings will be used to examine how joint motion and muscle activation change over the kicking movement. The study is expected to involve minimal risk, similar to routine sports testing. Possible discomforts include temporary muscle fatigue or mild soreness. Participants may not receive direct benefit, but the findings may inform training and injury-prevention strategies for taekwondo athletes. All collected data will be kept confidential and analyzed without personal identifiers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy taekwondo athletes currently training and actively participating in taekwondo.
* Able and willing to provide written informed consent (and assent with parental/guardian consent for minors, if applicable).
* Assigned to either the elite group or the youth group based on competition level and/or age category as defined in the study protocol.

Exclusion Criteria:

* Current pain, acute injury, or musculoskeletal disorder affecting the lower limbs or trunk that could influence kicking performance.
* Any injury or illness within the past 3 months that limited full training participation.
* Neurological, cardiovascular, or other medical condition that may make vigorous sport-specific testing unsafe.

Ages: 14 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Healthy taekwondo athletes recruited from local training centers/teams will be enrolled and categorized into an elite group and a youth group. Participants will attend a single laboratory visit to perform standardized roundhouse kick trials while lower-limb biomechanics are measured using motion analysis, force platforms, and surface electromyography.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Lower-Limb Joint Angles During the Taekwondo Roundhouse Kick | Day 1
  Time-series hip, knee, and ankle joint angles (degrees) during standardized roundhouse kick trials. Waveform-based analyses (including FPCA) will compare elite and youth athletes.
Lower-Limb Net Joint Moments During the Taekwondo Roundhouse Kick | Day 1
  Time-series net joint moments at the hip, knee, and ankle (Nm or normalized as Nm/kg) during standardized roundhouse kick trials. Waveform-based analyses (including FPCA) will compare groups.
Ground Reaction Forces During the Taekwondo Roundhouse Kick | Day 1
  Time-series ground reaction forces (N or normalized as N/body weight) collected from force platforms during kick trials (e.g., vertical/anterior-posterior/medial-lateral components). Group comparisons will use waveform-based analyses (including FPCA).
Surface EMG Amplitude Measures During the Taekwondo Roundhouse Kick | Day 1
  Surface EMG from selected lower-limb muscles recorded during kick trials. EMG amplitude outcomes include root mean square (RMS, µV) and integrated EMG (iEMG, µV·s), calculated over pre-specified phases of the kick. Comparisons will be made between elite and youth athletes.

CONTACTS AND LOCATIONS:
Locations (1):
- Sports Biomechanics Laboratory, Yantai, Shandong, China

IPD SHARING:
Plan to Share IPD: No